CLINICAL TRIAL: NCT06309381
Title: Rebound Pain After Outpatient Orthopaedic Foot Surgery Under Popliteal Sciatic Nerve Block: Influence of Sensory Block Duration. An Observational Study.
Brief Title: Influence of Sensory Block Duration on Rebound Pain After Outpatient Foot Surgery Under Popliteal Sciatic Nerve Block.
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Javier Barrio, MD, PhD, Hospital Universitario Doctor Peset
Other Study IDs: CEIm2.23
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Rebound Pain; Sciatic Nerve Block; Foot Surgery; Outpatient Surgery
Keywords: Acute Pain; Pain, Postoperative; Rebound pain; Sciatic Nerve Block; Orthopedic Procedures; Foot surgery; Outpatient Surgery
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rebound pain after surgeries under peripheral nerve block is defined as the appearance of severe acute postoperative pain after regression of the sensory block. The incidence of this condition can reach up to 40-50% in patients undergoing ambulatory surgeries. Rebound pain represents a clinically significant issue that may outweigh the benefits of regional anaesthesia. This is particularly significant for painful outpatient surgeries, where inadequately managed pain can result in distress, potentially affecting patient satisfaction and recovery. It may also lead to unplanned utilization of healthcare resources or readmissions.

Orthopaedic foot surgery is a prevalent outpatient surgery, potentially painful, where rebound may be a difficult challenge. However, to date, prospective studies focusing specifically on rebound pain in outpatient foot surgery are limited. Identifying conditions associated with rebound pain or at-risk patients could facilitate the development of preventive and treatment strategies, thereby enhancing pain management or relief. Younger age, female sex and bone surgery are non-modifiable factors associated with severe rebound pain. Perioperative intravenous dexamethasone has been identified as a modifiable independent risk factor associated with a reduced incidence of rebound pain. Regarding anaesthetic factors, the duration of the peripheral block has been proposed as a potentially modifiable factor influencing rebound pain; however, current evidence does not support this hypothesis.

The goal of this prospective observational study is to evaluate the incidence of rebound pain specifically in outpatient orthopaedic foot surgery involving bone under popliteal sciatic nerve block and to assess the possible association between sensory block duration and the incidence of rebound pain.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years old), ASA physical status 1 to 3, scheduled for elective outpatient orthopaedic foot surgery involving bone under popliteal sciatic nerve block.

Exclusion Criteria:

* age younger than 18 years, ASA physical status greater than 3, surgery not performed under popliteal sciatic nerve block or cases of failed sciatic nerve block, patients with type-1 diabetes or those under treatment for chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years old), ASA physical status class 1 to 3, scheduled for elective outpatient orthopaedic foot surgery involving bone under popliteal sciatic nerve block.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of rebound pain. | Up to 72 hours.
  Rebound pain is defined as the appearance of severe acute postoperative pain (numerical rating scale (NRS) ≥7) after regression of the sensory block of the sciatic nerve block.
  The highest self-reported NRS pain score after the block wears off and NRS pain scores at 24 hours, 48 hours and 72 hours (if necessary) after the block will be recorded.
Sensory block duration of the sciatic nerve block. | Up to 72 hours.
  Sensory block duration is defined as the time (hours) from block establishment to the appearance of pain at the surgical site.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Barrio, MD, PhD, Principal Investigator — Hospital Universitario Doctor Peset
Locations (1):
- Av. de Gaspar Aguilar, 90, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No